CLINICAL TRIAL: NCT05486559
Title: ECMO-Free Trial: A Multicenter Randomized Controlled Trial
Brief Title: The ECMO-Free Trial
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Whitney Gannon, Acute Care Nurse Practitioner, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 220733
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Extracorporeal Membrane Oxygenation Complication

STUDY DESIGN:
Intervention Model Description: Open-label, parallel-group, randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The ECMO-free Protocol group (Experimental): For patients assigned to the ECMO-free protocol group, the study personnel will perform the ECMO-free protocol daily from enrollment until the first of death or ECMO decannulation; results will be recorded and shared with the treatment team. Final decisions regarding decannulation will be made by treating clinicians who are aware of the results of daily ECMO-free protocolized assessments.
  Interventions: Other: ECMO-free protocol
- The Usual Care Group (Active Comparator): For patients assigned to the usual care group, ECMO weaning and assessments of readiness for ECMO decannulation will be at the discretion of treating clinicians.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: ECMO-free protocol — All patients randomized to the ECMO-Free Protocol Group will receive a protocolized daily assessment of readiness for liberation from VV-ECMO, which will be initiated between 6:00 AM local time and 10:00 AM local time. If the patient is enrolled after 10:00 AM local time the ECMO-free protocol will begin the following calendar day.
  The ECMO-Free Protocol is a 3-step process of assessing readiness for liberation from VV-ECMO: a safety screen (Phase 1: ECMO-Free Safety Screen), titration of the non-ECMO fraction of inspired oxygen (Phase 2: Non-ECMO respiratory support titration), and a trial of cessation of sweep gas flow (Phase 3: ECMO-Free Trial).
  Arms: The ECMO-free Protocol group
Other: Usual Care — All patients randomized to the Usual Care Group will undergo assessments of readiness for liberation, weaning, and decannulation at the discretion of the treatment team.
  Arms: The Usual Care Group

SUMMARY:
Decannulation from venovenous extracorporeal membrane oxygenation (VV-ECMO) at the earliest and safest time would be expected to improve outcomes and reduce cost. Daily assessments for readiness to liberate from therapies have demonstrated success in other realms of critical care. A recent single-center study demonstrated that a protocolized daily assessment of readiness for liberation from VV-ECMO was feasible and did not raise any major safety concerns, but the effect of this protocolized daily assessment on clinical outcomes remains unclear. Further, the manner in which ECMO is provided, weaned, and discontinued varies significantly between centers, raising persistent concerns regarding widespread adoption of protocolized daily assessment of readiness for liberation from VV-ECMO. Data from large a randomized controlled trial is needed to compare the effects of a protocolized daily assessment of readiness for liberation from VV-ECMO versus usual care on duration of ECMO support and other clinical outcomes.

DETAILED DESCRIPTION:
Complication rates, economic consequences, and resource limitations associated with the use of venovenous ECMO (VV-ECMO) are widely recognized. Decannulation at the earliest and safest possible time would be expected to improve clinical outcomes, reduce cost, and optimize resource allocation. Yet, there are no data comparing weaning strategies for decannulation from VV-ECMO, and there is significant variation between centers in approaches to weaning VV-ECMO.

Current approaches to weaning VV-ECMO generally rely on clinicians to identify signs of lung recovery and initiate incremental reductions in blood flow rate, fraction of delivered oxygen (FdO2), and sweep gas flow rate4-6. This approach has been previously outlined in guidelines distributed by the Extracorporeal Life Support Organization, expert opinion, and in small descriptive studies, though little data exist to support this strategy. Further, these approaches run counter to the large body of literature for assessing readiness for "liberation" from sedation and mechanical ventilation in which incremental reductions (weaning) have repeatedly been shown to be inferior to protocolized daily assessments (spontaneous awakening trials and spontaneous breathing trials7-11).

Prior data suggest that clinicians underestimate readiness for liberation from organ support and suggest that protocols to identify readiness for liberation are superior to clinician judgement9,11. Compared to incremental weaning, spontaneous awakening trials and spontaneous breathing trials have been shown to dramatically shorten the duration of support, reduce intensive care costs, and improve outcomes7-13. Until recently, this approach to liberating patients from a therapy had not been applied to ECMO. Our groups recently conducted a 26-patient, prospective, single-arm, safety and feasibility study to develop and refine a protocol for daily assessment of readiness to liberate from VV-ECMO at a single center14. The results of this study, published in CHEST, suggested that a protocolized daily assessment of readiness for liberation from VV-ECMO is feasible and safe. Further, the median time from first passed trial to decannulation was 2 days, suggesting that a daily protocolized assessment might identify candidates for decannulation earlier than occurs in usual care. However, as a single-arm feasibility study, the prior study was insufficient to determine whether dedicating resources to a protocolized daily assessment of readiness to liberate from VV-ECMO affects patient outcomes. Further, the manner in which ECMO is provided, weaned, and discontinued varies significantly between centers, raising persistent concerns regarding the feasibility of widespread adoption of protocolized daily assessment of readiness for liberation from VV-ECMO.

Additional data from a large, multi-center randomized controlled trial are needed to compare the effects of a protocolized daily assessment of readiness for liberation from VV-ECMO versus usual care on duration of ECMO support, measures of unsafe liberation, and other clinical outcomes.

Primary aim: Compare the effects of a protocolized daily assessment of readiness for liberation from VV-ECMO (ECMO-free protocol) versus liberation strategy directed by the clinical team (usual care) on time to successful decannulation via a large multi-site randomized controlled trial.

Secondary aim: To compare the effect of a once daily protocolized assessment of readiness to liberate from ECMO (ECMO-free protocol) versus a liberation strategy directed by the clinical team (usual care) on the number of days alive and free of ECMO by day 60 (ECMO-free days).

To address these aims, we propose a multi-center, open-label, parallel-group, randomized controlled trial comparing a protocolized daily assessment of readiness for liberation from VV-ECMO (ECMO-free protocol) to usual care. All patients who receive VV-ECMO in a participating unit of an adult hospital and meet all inclusion criteria and no exclusion criteria will be eligible for participation. Eligible participants or surrogate decision makers will be approached for consent. Following documentation of written informed consent, patients will be enrolled and randomly assigned to receive the ECMO-free protocol or usual care. The study will control VV-ECMO weaning strategy until the first of decannulation or death. All other decisions regarding critical care support, interventional therapies, and medical treatment will remain at the discretion of the treating physician and consulting teams.

ELIGIBILITY:
Inclusion Criteria:

* Patient receiving VV-ECMO
* Patient is located in a participating unit of an adult hospital

Exclusion Criteria:

* Patient is pregnant
* Patient is a prisoner
* Patient is < 18 years old
* Participant is receiving ECMO as bridge to transplant
* Participant is receiving a hybrid configuration that includes an arterial cannula
* Patient has received VV-ECMO for > 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2022-09-07 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Time to successful discontinuation of ECMO | From randomization to time of hospital discharge or until day 60.
  The primary outcome will be the time (in days) from randomization (time zero) until the time of the final successful discontinuation of ECMO. Discontinuation of ECMO will be considered to be successful if a patient undergoes decannulation and survives without ECMO until day 60. For patients who are decannulated and subsequently experience recannulation, the time of successful discontinuation of ECMO will be based on the final decannulation. Data collection will cease at the time of hospital discharge or day 60.

SECONDARY OUTCOMES:
ECMO-free days to day 60 | From randomization to death or hospital discharge through day 60.
  The number of days alive and free of ECMO to day 60 (ECMO-free days) will be calculated as 60 minus the number of calendar days from randomization to final decannulation. Patients receiving ECMO at day 60 will receive a value of "0". Patients who die before day 60 or hospital discharge will receive a value of "0".

OTHER OUTCOMES:
Unsafe discontinuation of ECMO | From randomization to 48 hours after decannulation.
  Unsafe liberation will be defined according to a previously published definition.1 A patient will be classified as having experienced unsafe discontinuation of ECMO if he or she experiences any of the following within 48 hours of decannulation: VV-ECMO recannulation, sustained (> 4 hours) escalation of mechanical ventilation (change from a partially assisted mode to controlled MV, or dynamic driving pressure greater than or equal to 16 and delta change from previous setting of greater than or equal to 5 cm H2O, or increase in FiO2 to > 80%), use of rescue therapies (i.e. new need for paralysis and deep sedation, or inhaled pulmonary vasodilators, or high frequency oscillatory ventilation, or new worsening hemodynamics requiring addition of any vasoactive agents with no evidence of sepsis or hypovolemia).
Recannulation within 30 days of decannulation | From decannulation until 30 days after decannulation.
  Reinstituting ECMO support within 30 days of discontinuation.
Survival to decannulation | From randomization to until the date of death or the date of decannulation, whichever came first, through day 60.
  Alive at time of decannulation
Respiratory support-free days to day 60 | From randomization to the date of death or discharge, whichever came first, through day 60.
  Number of days free of respiratory support between randomization and day 60.
ICU-free days to day 60 | From randomization to the date of death or discharge, whichever came first, through day 60.
  Number of days alive and not in the ICU between randomization and day 60.
Ventilator-free days to day 60 | From randomization to the date of death or discharge, whichever came first, through day 60.
  Number of days alive and free from mechanical ventilation between randomization and day 60.
Hospital-free days to day 60 | From randomization to the date of death or discharge, whichever came first, through day 60.
  Number of days alive and not in the hospital between randomization and day 60.
60-day in-hospital mortality | From randomization to the date of death or discharge, whichever came first, through day 60.
  Death prior to hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Casey, MD, MSc, Study Director — Vanderbilt University Medical Center
Locations (8):
- United States (7):
  - UC San Diego Health, San Diego, California
  - Stanford University, Stanford, California
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - University of Utah Health, Salt Lake City, Utah
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Al-Fares AA, Ferguson ND, Ma J, Cypel M, Keshavjee S, Fan E, Del Sorbo L. Achieving Safe Liberation During Weaning From VV-ECMO in Patients With Severe ARDS: The Role of Tidal Volume and Inspiratory Effort. Chest. 2021 Nov;160(5):1704-1713. doi: 10.1016/j.chest.2021.05.068. Epub 2021 Jun 21. PMID 34166645
- [Background] Peek GJ, Mugford M, Tiruvoipati R, Wilson A, Allen E, Thalanany MM, Hibbert CL, Truesdale A, Clemens F, Cooper N, Firmin RK, Elbourne D; CESAR trial collaboration. Efficacy and economic assessment of conventional ventilatory support versus extracorporeal membrane oxygenation for severe adult respiratory failure (CESAR): a multicentre randomised controlled trial. Lancet. 2009 Oct 17;374(9698):1351-63. doi: 10.1016/S0140-6736(09)61069-2. Epub 2009 Sep 15. PMID 19762075
- [Background] Brodie D, Slutsky AS, Combes A. Extracorporeal Life Support for Adults With Respiratory Failure and Related Indications: A Review. JAMA. 2019 Aug 13;322(6):557-568. doi: 10.1001/jama.2019.9302. PMID 31408142
- [Background] Broman LM, Malfertheiner MV, Montisci A, Pappalardo F. Weaning from veno-venous extracorporeal membrane oxygenation: how I do it. J Thorac Dis. 2018 Mar;10(Suppl 5):S692-S697. doi: 10.21037/jtd.2017.09.95. PMID 29732188
- [Background] Vasques F, Romitti F, Gattinoni L, Camporota L. How I wean patients from veno-venous extra-corporeal membrane oxygenation. Crit Care. 2019 Sep 18;23(1):316. doi: 10.1186/s13054-019-2592-5. No abstract available. PMID 31533848
- [Background] Grant AA, Hart VJ, Lineen EB, Badiye A, Byers PM, Patel A, Vianna R, Koerner MM, El Banayosy A, Loebe M, Ghodsizad A. A Weaning Protocol for Venovenous Extracorporeal Membrane Oxygenation With a Review of the Literature. Artif Organs. 2018 Jun;42(6):605-610. doi: 10.1111/aor.13087. Epub 2018 Jan 18. PMID 29344952
- [Background] Kress JP, Pohlman AS, O'Connor MF, Hall JB. Daily interruption of sedative infusions in critically ill patients undergoing mechanical ventilation. N Engl J Med. 2000 May 18;342(20):1471-7. doi: 10.1056/NEJM200005183422002. PMID 10816184
- [Background] Brook AD, Ahrens TS, Schaiff R, Prentice D, Sherman G, Shannon W, Kollef MH. Effect of a nursing-implemented sedation protocol on the duration of mechanical ventilation. Crit Care Med. 1999 Dec;27(12):2609-15. doi: 10.1097/00003246-199912000-00001. PMID 10628598
- [Background] Girard TD, Kress JP, Fuchs BD, Thomason JW, Schweickert WD, Pun BT, Taichman DB, Dunn JG, Pohlman AS, Kinniry PA, Jackson JC, Canonico AE, Light RW, Shintani AK, Thompson JL, Gordon SM, Hall JB, Dittus RS, Bernard GR, Ely EW. Efficacy and safety of a paired sedation and ventilator weaning protocol for mechanically ventilated patients in intensive care (Awakening and Breathing Controlled trial): a randomised controlled trial. Lancet. 2008 Jan 12;371(9607):126-34. doi: 10.1016/S0140-6736(08)60105-1. PMID 18191684
- [Background] Ely EW, Baker AM, Dunagan DP, Burke HL, Smith AC, Kelly PT, Johnson MM, Browder RW, Bowton DL, Haponik EF. Effect on the duration of mechanical ventilation of identifying patients capable of breathing spontaneously. N Engl J Med. 1996 Dec 19;335(25):1864-9. doi: 10.1056/NEJM199612193352502. PMID 8948561
- [Background] Ely EW, Meade MO, Haponik EF, Kollef MH, Cook DJ, Guyatt GH, Stoller JK. Mechanical ventilator weaning protocols driven by nonphysician health-care professionals: evidence-based clinical practice guidelines. Chest. 2001 Dec;120(6 Suppl):454S-63S. doi: 10.1378/chest.120.6_suppl.454s. PMID 11742965
- [Background] Brochard L, Rauss A, Benito S, Conti G, Mancebo J, Rekik N, Gasparetto A, Lemaire F. Comparison of three methods of gradual withdrawal from ventilatory support during weaning from mechanical ventilation. Am J Respir Crit Care Med. 1994 Oct;150(4):896-903. doi: 10.1164/ajrccm.150.4.7921460.
- [Background] Esteban A, Frutos F, Tobin MJ, Alia I, Solsona JF, Valverdu I, Fernandez R, de la Cal MA, Benito S, Tomas R, et al. A comparison of four methods of weaning patients from mechanical ventilation. Spanish Lung Failure Collaborative Group. N Engl J Med. 1995 Feb 9;332(6):345-50. doi: 10.1056/NEJM199502093320601. PMID 7823995
- [Background] Gannon WD, Stokes JW, Bloom S, Sherrill W, Bacchetta M, Rice TW, Semler MW, Casey JD. Safety and Feasibility of a Protocolized Daily Assessment of Readiness for Liberation From Venovenous Extracorporeal Membrane Oxygenation. Chest. 2021 Nov;160(5):1693-1703. doi: 10.1016/j.chest.2021.05.066. Epub 2021 Jun 21. PMID 34166644
- [Derived] Gannon WD, Teijeiro-Paradis R, Prekker ME, Vogelsong MA, Schwartz GS, Odish MF, Nickel NP, Bloom SL, Hansen SJ, Fielding-Singh V, Blough B, Owens RL, Valles R, Adkisson WS, Alvis BD, Bacchetta M, Ford DJ, Gaudio SC, Jelly CA, Landsperger JS, Lingle K, Noblit CC, Rice TW, Del Sorbo L, Stokes JW, Stollings JL, Van Winkle G, Wang L, Imhoff B, Shotwell MS, Fan E, Semler MW, Casey JD; ECMO-Free Investigators and the Pragmatic Critical Care Research Group. Protocol and Statistical Analysis Plan for the ECMO-Free Trial: A Multicenter Randomized Controlled Trial. medRxiv [Preprint]. 2025 Dec 2:2025.12.01.25341410. doi: 10.64898/2025.12.01.25341410. PMID 41404271